CLINICAL TRIAL: NCT07269925
Title: Impact of Different Electrical Frequencies Used in Percutaneous Neuromodulation on Muscle Strength and Pressure Pain Thresholds
Acronym: PENS-DOSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, JUAN ANTONIO VALERA CALERO, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UComplutenseMadrid-PENS
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Shoulder Pain
Keywords: Percutaneous electrical nerve stimulation; Strength; Pain pressure thresholds
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blinded, Placebo-Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Frequency PENS (Experimental): Participants will receive a single session of PENS setting 2 Hz frequency, 250 µs pulse width, 10 minutes duration, with an intensity (mA) sufficient to elicit a visible motor response while remaining comfortable for the patient.
  Interventions: Other: Percutaneous electrical nerve stimulation: Low frequency
- High Frequency PENS (Experimental): Participants will receive a single session of PENS setting 100 Hz frequency, 250 µs pulse width, 5-second stimulation followed by 55-second rest, with an intensity (mA) sufficient to elicit a visible motor response while remaining comfortable for the patient and repeated five times.
  Interventions: Other: Percutaneous electrical nerve stimulation: High frequency

INTERVENTIONS:
Other: Percutaneous electrical nerve stimulation: High frequency — A single PENS session will be applied under ultrasound guidance using sterile, single-use filiform needles placed in the suprascapular and axillary nerves and connected to an electrostimulator APSe4 (Agupunt, Barcelona).
  Dosage will be: 100 Hz frequency, 250 µs pulse width, 5-second stimulation followed by 55-second rest, repeated five times
  Arms: High Frequency PENS
Other: Percutaneous electrical nerve stimulation: Low frequency — A single PENS session will be applied under ultrasound guidance using sterile, single-use filiform needles placed in the suprascapular and axillary nerves and connected to an electrostimulator APSe4 (Agupunt, Barcelona). Dosage will be: 2 Hz frequency, 250 µs pulse width, 10 minutes duration, with an intensity (mA) sufficient to elicit a visible motor response while remaining comfortable for the patient.
  Arms: Low Frequency PENS

SUMMARY:
Percutaneous electrical nerve stimulation (PENS) involves delivering electrical currents through fine filiform needles inserted near tissues such as muscles, ligaments, or nerves. It has been explored for various chronic pain conditions affecting the cervical and lumbar spine, as well as the upper and lower limbs. Despite its growing clinical use, the overall quality of evidence supporting PENS for chronic musculoskeletal pain remains limited. Most studies have applied the technique directly over nerve structures, and while some reviews have shown greater pain reduction compared to transcutaneous electrical nerve stimulation (TENS), the superiority of PENS has not been conclusively demonstrated. Research specifically examining its application on nerve tissues, particularly in the upper limbs, remains scarce. Some preliminary and single-case studies have reported improvements in pain and disability following PENS directed at the radial nerve, but these findings are limited by small sample sizes and the absence of control groups. The physiological mechanisms underlying PENS are still not fully understood, though both peripheral and central processes are believed to be involved. Evidence suggests that PENS can reduce local sensitivity to pressure pain through peripheral mechanisms and may also enhance descending inhibitory control by activating conditioned pain modulation at the central level. However, further studies are necessary to clarify these effects.

Since to date, limited research has specifically examined the optimal PENS dosage, the present study aimed to compare two PENS dosage for improving muscle strength and pain pressure thresholds.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one latent myofascial trigger point (MTrP) in the infraspinatus muscle, identified according to the most recent Delphi consensus criteria.
* Ability to read, understand, and sign the written informed consent form.

Exclusion Criteria:

* Current pharmacological treatment that may affect muscle tone.
* History of shoulder or spinal surgery.
* Traumatic disorders such as whiplash-associated injuries, dislocations, or fractures.
* Neuropathies, including radiculopathies or myelopathies.
* Severe medical conditions (e.g., tumors, fractures, neurological or systemic diseases).
* Clinically relevant asymmetries.
* Generalized musculoskeletal conditions such as fibromyalgia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | Baseline
  Shoulder external rotator strength will be assessed using a handheld dynamometer (TruStrength, Hawkin Dynamics, USA), previously validated for measuring isometric muscle contraction strength. Participants will perform a standardized isometric external rotation test in a seated position with the elbow flexed at 90°.
Muscle strength | Post-intervention (10 minutes)
  Shoulder external rotator strength will be assessed using a handheld dynamometer (TruStrength, Hawkin Dynamics, USA), previously validated for measuring isometric muscle contraction strength. Participants will perform a standardized isometric external rotation test in a seated position with the elbow flexed at 90°.

SECONDARY OUTCOMES:
Pain Pressure Thresholds - Latent MTrP | Baseline
  The assessment of pressure pain thresholds (PPT) at the myofascial trigger point (MTrP) will be evaluated three times at each measurement site using a analog algometer, applying a pressure rate of approximately 5 N/s.
Pain Pressure Thresholds - Latent MTrP | Post-intervention (10 minutes)
  The assessment of pressure pain thresholds (PPT) at the myofascial trigger point (MTrP) will be evaluated three times at each measurement site using a analog algometer, applying a pressure rate of approximately 5 N/s.
Pain Pressure Thresholds - Tibialis anterior | Baseline
  The assessment of pressure pain thresholds (PPT) at a distal location (Tibia's anterior) will be evaluated three times at each measurement site using a analog algometer, applying a pressure rate of approximately 5 N/s.
Pain Pressure Thresholds - Tibialis anterior | Post-intervention (10 minutes)
  The assessment of pressure pain thresholds (PPT) at a distal location (Tibia's anterior) will be evaluated three times at each measurement site using a analog algometer, applying a pressure rate of approximately 5 N/s.

CONTACTS AND LOCATIONS:
Locations (1):
- ATMIS, Krakow, Poland, Poland

IPD SHARING:
Plan to Share IPD: Undecided